CLINICAL TRIAL: NCT03318406
Title: Post-Market Registry for Patients With Emphysema Treated With BTVA
Brief Title: Post-Market BTVA Registry
Status: Recruiting | Type: Observational
Sponsor: Uptake Medical Technology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP-2410
Record Dates: First submitted 2017-10-13; First posted 2017-10-23 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Emphysema or COPD
Keywords: registry; vapor ablation; InterVapor; BTVA
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- BTVA treated patients: Patients with heterogeneous upper lobe emphysema undergoing Bronchoscopic Thermal Vapor Ablation treatment
  Interventions: Device: Bronchoscopic Thermal Vapor Ablation

INTERVENTIONS:
Device: Bronchoscopic Thermal Vapor Ablation — Bronchoscopic vapor delivery to airway segment(s) targeted for treatment
  Other Names: BTVA; InterVapor

SUMMARY:
Bronchoscopic thermal vapor ablation using Uptake Medical Technology Inc.'s InterVapor System is indicated for treatment of patients with heterogeneous upper lobe emphysema. This study is a retrospective and prospective, observational, multi-center, post-market registry of patients prescribed InterVapor. The primary objective of the Registry is to describe the long-term impact of InterVapor treatment on patient quality of life (QOL) in a real-world setting. After InterVapor treatment, patients will be followed for 5 years as per the standard of care and safety and efficacy data (quality of life, pulmonary function, exercise capacity) collected as part of the registry.

DETAILED DESCRIPTION:
The BTVA Registry will enroll up to 300 patients with upper lobe predominant emphysema that are being treated with BTVA at sites located in the EU and other select geographies. Patients will be followed as per standard of care and the registry will collect follow-up data for five years following treatment. The follow up data collected will include pulmonary function measurements (spirometry, body plethysmography, and diffusing capacity for carbon monoxide), exercise capacity (six minute walk test), imaging findings (chest x-ray and CT), and a quality of life questionnaire (SGRQ-C). All serious and non-serious adverse events will also be collected for the duration of the study in order to assess safety. Serious adverse events will be adjudicated by an independent medical monitor in order to establish relatedness to the InterVapor device and procedure.

Descriptive statistics will be used to summarize all safety and effectiveness data. There is no predefined hypothesis regarding the magnitude of effectiveness of InterVapor or the incidence of specific safety outcomes.

Monitoring of the registry study will be undertaken as a continuous process to ensure that high-quality data are obtained and to ensure compliance with registry procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will have heterogeneous emphysema, as evidenced by high-resolution computed tomography (HRCT) demonstrating a heterogeneity index > or equal to 1.2 in at least one segment to be treated
2. Patients must be > or equal to 18 years of age
3. Patients are required to provide informed consent prior to inclusion in the Registry

Exclusion Criteria:

1. FEV1 < 20% predicted
2. DLCO < 20% predicted
3. Inability to walk > 140 meters in 6 minutes (6MWD) following optimized medical management
4. Unstable COPD (any of the following):

   1. > 3 COPD related hospitalizations requiring antibiotics in past 12 months
   2. COPD related hospitalization in past 3 months
   3. daily use of systemic steroids, i.e. > 5 mg prednisolone
5. Concomitant illnesses or medications that would pose a significant increased risk for complications following treatment with InterVapor. Examples of particular relevance include: immune system disorders, immunosuppressant medications of clinical relevance, bleeding disorders and unstable cardiovascular conditions, history of asthma or alpha-1 antitrypsin deficiency
6. Newly prescribed morphine derivatives within the last 4 weeks
7. Pregnant or breastfeeding
8. Highly diseased lower lobes (tissue to air ratio of <11%)
9. Bacterial infection or symptoms indicative of active infection (i.e., fever, elevated white blood cell count)
10. Presence of single large bulla (defined as > 1/3 volume of lobe) or a paraseptal distribution of emphysema in the treated lobe
11. Recent respiratory infections or COPD exacerbation in preceding 6 weeks -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with upper lobe predominant emphysema being evaluated for possible InterVapor treatment will be considered for enrollment in the Registry
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-03-22 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life | Baseline to 24 months
  Change in Quality of Life score as assessed by the SGRQ-C questionnaire

SECONDARY OUTCOMES:
Serious Adverse Events | 6 and 12 months
  procedure and device related serious adverse events, major medical complications
Change in FEV1 | Baseline to 12 months
  Change in Forced Expired Volume in 1 second
Change in FVC | Baseline to 12 months
  Change in Forced Vital Capacity
Change in TLC | Baseline to 12 months
  Change in Total Lung Capacity
Change in RV | Baseline to 12 months
  Change in Residual Volume
Change in DLCO | Baseline to 12 months
  Change in Diffusing capacity of the lung for carbon monoxide
Exercise Tolerance | Baseline to 12 months
  Change in six minute walk distance
Lung volume reduction | Baseline to 6 months
  change in lung volume assessed by CT

CONTACTS AND LOCATIONS:
Overall Officials: Felix Herth, MD, PhD, Principal Investigator — Thoraxklinik University of Heidelberg
Locations (20):
- Krankenhaus Nord - Klinik Floridsdorf, Vienna, Austria
- Germany (13):
  - Sozialstiftung Bamberg, Klinikum am Bruderwald, Bamberg
  - DRK Kliniken Berlin / Mitte, Berlin
  - FORSCHUNGSINSTITUT Havelhöhe gGmbH, Berlin
  - Ruhrlandklinik - Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Asklepios Fachkliniken München-Gauting, Gauting
  - Martin-Luther-Universität Halle-Wittenberg (Saale), Halle
  - Thoraxklinik Heidelberg, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Lungenfachklinik Immenhausen, Immenhausen
  - Krankenhaus Martha-Maria München, München
  - Klinikum Nürnberg Nord, Nuremberg
  - Krankenhaus vom Roten Kreuz Bad Cannstatt GmbH, Stuttgart
  - Klinik Schillerhöhe, Stuttgart
- Switzerland (6):
  - Kantonsspital Aarau AG, Aarau
  - University Hospital Basel, Basel
  - Lungen-und Schlafzentrum am Lindenhofspital AG, Bern, Bern
  - Kantonsspital St.Gallen, Sankt Gallen
  - LungenZentrum Hirslanden, Zurich
  - Universitäts Spital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No